CLINICAL TRIAL: NCT05862246
Title: Is There an Association Between Gastrocnemius Tightness and Foot- and Legpain in Children?
Brief Title: Gastrocnemius Tightness and Foot Pain in Children
Status: Recruiting | Type: Observational
Sponsor: St. Olavs Hospital (Other)
Collaborators: National Taiwan Normal University (Other)
Responsible Party: Sponsor
Other Study IDs: 526706
Record Dates: First submitted 2023-05-08; First posted 2023-05-17 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Child Development; Gastrocnemius Equinus
MeSH Terms: interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children with pain: These are children referred with fot and leg pain. Following outcomes will be measured on all included children:
  Silvferskiölds test Height Weight Gender Age PROM child: Oxford Ankle and Foot Questionnaire for children PROM parent: Oxford Ankle and Foot Questionnaire for parents FPS pain scoring over 1 week
  Interventions: Other: Clinical examination
- Control group children without pain: Following outcomes will be measured on all included children in control group:
  Silvferskiölds test Height Weight Gender Age
  Interventions: Other: Clinical examination

INTERVENTIONS:
Other: Clinical examination — No intervention, only clinical examination

SUMMARY:
Foot and leg pain among otherwise healthy children is a common reason for referral to our pediatric orthopaedics outpatient clinic. The pain is often intermittent and transient, but for some the pain is more dominating and has an impact on the child and families. Children grown and have normal anatomical variations such as in-toeing, out-toeing, hypermobility, flatfeet, knock knees etc. Assessing such normal variants is a major part of pediatric orthopaedic practice, and a common finding is a positive Silvferskiöld test, indicating gastrocnemius tightness. This is when dorsiflexion of the ankle is limited with extended knee, compared to flexed knee. We do not know if this is a more frequent finding among children with foot and leg pain. There is however evidence that adults with painful foot conditions often have gastrocnemius tightness.

This project will investigate for gastrocnemius tightness in otherwise healthy children referred to our pediatric orthopaedic outpatient clinic with foot and leg pain, and compare results with a similar control group of children without pain. The aim is to investigate if there is an association, and how pain and tightness develops over time. The knowledge from this project will enable us to develop new treatment strategies to this patient group, where current evidence based recommendations are few.

ELIGIBILITY:
Inclusion Criteria:

* Otherwise healthy children referred to pediatric orthopaedic outpatient clinic with foot and/or leg pain with a normal leg function

Exclusion Criteria:

* Patients with foot conditions, general medical conditions affecting the foot or clinical findings indicating a need for further investigation for a diagnosis. Such as:

Foot deformities (cavo-varus foot, clubfoot) Tarsal coalitions Neuro-orthopedic conditions (CP, MMC) Fracture sequelae Infections and tumour

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children referred to pediatric orthopaedic outpatients clinic from a family doctor
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-05-09 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Silvferskiölds test | 2 years
  Clinical measurement of gastrocnemius tightness

CONTACTS AND LOCATIONS:
Overall Officials: Håkon Langvatn, Principal Investigator — St. Olavs Hospital
Locations (1):
- St Olavs hospital, Trondheim, Norway